CLINICAL TRIAL: NCT06059898
Title: A Randomized Clinical Study Comparing the Bioresorbable Magnesium NOVAMag® Membrane With the Collagen Jason® Membrane in Patients Requiring Guided Bone Regeneration
Brief Title: Magnesium NOVAMag® Membrane vs. Collagen Jason® Membrane in Patients Requiring Guided Bone Regeneration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Botiss Medical AG (Other)
Collaborators: CONVIDIA clinical research GmbH (Unknown); Botiss Biomaterials GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NM-MEM-01
Record Dates: First submitted 2023-09-04; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Guided Bone Regeneration (GBR); Ridge Augmentation; Periodontal Bone Defect
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NOVAMag membrane (Experimental): GBR procedure / membrane placement
  Interventions: Device: GBR surgery including membrane placement; Procedure: Biopsy
- Jason membrane (Active Comparator): GBR procedure / membrane placement
  Interventions: Device: GBR surgery including membrane placement; Procedure: Biopsy

INTERVENTIONS:
Device: GBR surgery including membrane placement — After the application of local anesthesia, an incision of the mucosa will be performed and the flap will be elevated. The flap closure line should not be directly over the defect, but away from the defect site to prevent wound dehiscence. The bony defect will be thoroughly cleaned and, in some cases, activated by drilling small holes in the cortical bone to increase blood flow into the bone graft. Bone substitute will be inserted, the membrane will be adapted and fixed, and the flap will be sutured
Procedure: Biopsy — After a healing period of 6 months, at the implantation site, a biopsy is taken from the site of dental implant insertion for further analysis of bone regeneration

SUMMARY:
The NOVAMag® membrane is a medical device approved in the EU, and is a completely resorbable and biodegradable metal membrane. This medical device is used in the treatment of bone defects in the oral cavity. The membrane ensures sufficient stability of the bone augmentation material and provides a barrier to the soft tissue. This enables new bone to form in the defect space and for the subsequent placement of dental implants. In this clinical trial, the NOVAMag® membrane is compared with the Jason® collagen membrane, another medical device for supporting bone regeneration, with the aim of demonstrating the non-inferiority in terms of radiographically measured volumetric bone gain of the NOVAMag® membrane to the comparator membrane.

DETAILED DESCRIPTION:
GBR is a well-established surgical procedure based on the use of tissue barriers to separate the void of hard tissue defects from overlying connective tissues, thus preventing the ingrowth of soft tissue into the defect site resulting in improved bone regeneration. GBR is used both with and without different bone graft materials, such as allografts, xenografts and synthetic substitute materials, which have shown comparable results to those obtained with autologous bone in localized horizontal defects.

The barrier membranes used in GBR can be produced from animal (bovine, porcine), human (allogenic) and synthetic biomaterials. Due to their origin, composition and manufacturing process, each biomaterial performs differently in the human body, with their own associated advantages and disadvantages.

Non-resorbable membranes (primarily made from PTFE [polytetrafluoroethylene] and titanium] can offer mechanical reinforcement to protect the defect void, as well as maintain a continuous barrier function until they are removed. The main disadvantage of these membranes is the necessity of a second surgical procedure for their removal.

In response to this disadvantage, resorbable membranes have been developed with porcine collagen membranes considering the standard product for use in GBR. These collagen membranes produce excellent biocompatible results, but they lack mechanical stability, especially for use in larger augmentation sites. To address the aforementioned issues of both the resorbable and non-resorbable membranes, botiss biomaterials GmbH has developed the NOVAMag® membrane, which has recently received CE approval. The NOVAMag® membrane is a resorbable, biodegradable magnesium membrane. The material properties of the pure magnesium membrane culminate into a design that has a mechanical stability not provided by other resorbable membranes. Despite being resorbable, the membrane maintains a separation of the soft and hard tissues until the bony defect has been repaired (data on file at botiss). The ability of membranes to resist collapse into the defect void and maintain space for the ingrowth of new bone is viewed as an important aspect for producing a successful regenerative outcome. This is most easily achieved by using a strong material that can resist the external pressures of the overlying soft tissue and the forces experienced during function. The risk of collapse tends to be higher for resorbable membranes due to inferior mechanical properties. Mechanical testing performed by botiss have proven that the magnesium membrane is self-supporting and substantially stronger than other resorbable collagen membranes. Therefore, the risk of collapse into the defect void, as reported for collagen membranes, could potentially be prevented by using the NOVAMag® membrane.

The aim of this randomized clinical study is to compare a bioresorbable magnesium NOVAMag® membrane with the collagen Jason® membrane in patients requiring guided bone regeneration.

ELIGIBILITY:
Inclusion Criteria:

1. Obtained informed consent from the patient, patients voluntarily signing the informed consent form before study related actions including patient's acceptance of the scheduled program of clinical and radiographic analysis
2. The patient shall be at least 18 years of age, male or female and have passed cessation of growth
3. Patients asking for more than one dental implant and presenting one site with a healed site (class h1i, h2i; h3i, v1i, c1i, h1e, h2e, h3e, Cologne Classification of Alveolar Ridge Defects (CCARD) requiring a GBR procedure prior to implant placement.
4. The teeth at the implant site must have been extracted or lost at least 8 weeks before the date of bone augmentation (volumetrically healed site)

Exclusion Criteria:

Systemic exclusion criteria

1. Major systemic diseases (e.g. recent myocardial infarction, cerebrovascular accident or valvular prosthesis surgery, a poorly stabilized diabetes mellitus, severe hypertension, severe peripheral artery occlusive disease, malignancies, autoimmune diseases, or kidney diseases, untreated or uncontrolled periodontal disease, uncontrolled drug or alcohol abuse, uncontrolled psychiatric disorders)
2. Acute infectious diseases
3. Immunocompromised patients
4. Serious disturbances of bone metabolism and/or serious bone diseases of endocrine etiology
5. Due to judgement of the principal investigator: Medical conditions requiring prolonged use of steroids and/or on-going treatment with gluco- and mineralocorticoids and with agents affecting calcium metabolism (e.g. calcitonin), and/or anti-coagulative therapy
6. Previous or current use of antiresorptive medication (e.g. bisphosphonates)
7. Previous oral / maxillofacial radiotherapy
8. Heavy smoker (definition: >10 cigarettes per day)
9. Currently pregnant or breastfeeding women
10. Health conditions, which do not permit the surgical treatment

Local exclusion criteria

1. Acute local inflammation or untreated periodontitis
2. Insufficient oral hygiene
3. Regenerative periodontal treatment necessary adjacent to the planned study site of interest
4. Mucosal diseases or oral white or ulcerative lesions (e.g. lichen planus, leukoplakia)
5. History of head and neck irradiation therapy
6. Severe bruxism or clenching or other destructive habits
7. Previous socket preservation, GBR or guided tissue regeneration (GTR) treatment at the implant site
8. Infections in tissue and adjacent tissue of the planned implantation site
9. Known hypersensitivity to any of the trace elements
10. Edentulous cases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-04-08 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Relative difference in bone volume between the groups at the augmentation site after GBR measured radiographically | Pre-treatment visit (T-1) to the clinical check up visit after five and a half months (T4)
  Mean volumetric increase in %

SECONDARY OUTCOMES:
Histomorphometric assessment of the differences in bone volume between the groups | T5: after a healing period of 6 months
  After 6 months a biopsy is taken from the site of dental implant insertion for further analysis. Undecalcified thin ground sections will be prepared. The following variables will be determined:
  * Bone volume per tissue volume in % (BV/TV)
  * New bone volume per tissue volume in % (nBV/TV)
  * Old bone volume per tissue volume in % (oBV/TV)
  * Total graft volume per tissue volume in % (GV/TV)
Evaluation of between group differences for the presence of side effects | At each follow-up visit: T1 (after 7-10 days), T2 (after 14 ± 3 days), T3 (after 1 month ± 4 days) and T5 (after 6 months ± 2 weeks)
  Presence or absence of side effects will be evaluated by the investigator during the scheduled follow-up appointments.
  Side effects to be assessed are:
  * Gas formation
  * Prickly feeling at surgery site (dysesthesia)
  * Redness/swelling
  * Bleeding
  * Wound dehiscence
  * Infection
  * Abscess/pus formation
Evaluation of between group differences for pain | At each follow-up visit: T1 (after 7-10 days), T2 (after 14 ± 3 days), T3 (after 1 month ± 4 days) and T5 (after 6 months ± 2 weeks)
  Pain will be self-assessed by the patients via a numerical rating scale (NRS) during the scheduled follow-up appointments. The scale has a measurement range of 0 to 10 (each inclusive). The higher the value, the more pain the patients experience.
Safety outcome measures | At T-1 (pre-treatment), T0 (= day 0 = day of surgery), T1 (after 7-10 days), T2 (after 14 ± 3 days), T3 (after 1 month ± 4 days), T5 (after 6 months ± 2 weeks), T6 (7-10 days after T5)
  The following Safety Endpoints will be evaluated by group at each visit:
  * Adverse events (AE) and Serious adverse events (SAEs)
  * Device related adverse events (adverse device effects (ADE)
  * Seriousness of device related adverse events (serious adverse device effect (SADE)
  * Device deficiency (DD)
Usability of the NOVAMag® membrane and its accessory products | At the end of the visit T0 [= day 0 = directly after GBR surgery]
  By completing a survey regarding the handling of the NOVAMag® membrane and its accessories by the investigator the usability will be evaluated.
Radiographic outcome measure: Changes in horizontal bone dimensions over time in mm. | At T-1 (pre-treatment) and T4 (5 and a half months ± 2 weeks)
  At T-1 and T4 a Cone Beam Computed Tomography (CBCT) is taken. CBCTs are compared and horizontal bone dimensions are measured at 2 mm, 4 mm, and 6 mm from the crest.
Radiographic outcome measure: Changes in vertical bone dimensions over time in mm. | At T-1 (pre-treatment) and T4 (5 and a half months ± 2 weeks)
  At T-1 and T4 a Cone Beam Computed Tomography (CBCT) is taken. CBCTs are compared and vertical bone dimensions are measured in mm.
Radiographic outcome measure: Bone quality assessment | T4 (after 5 and a half months ± 2 weeks)
  Bone quality assessment by evaluation of presence or absence of gas cavities by analysis of CBCT images after 6 months (only presence is reported from X-rays)

CONTACTS AND LOCATIONS:
Overall Officials: Werner Zechner, Prof. DDr., Principal Investigator — University of Vienna, Department of Oral Surgery, Austria
Locations (5):
- Austria (2):
  - Medical University of Graz Department of Dental Medicine and Oral Health, Graz
  - University of Vienna, Department of Oral Surgery, Vienna
- Copenhagen University Hospital, Department of Oral & Maxillofacial Surgery, Copenhagen, Denmark
- Italy (2):
  - Studio medico odontoiatrico Papi Stp Srl, Roma
  - Studio Tabanella, Roma

IPD SHARING:
Plan to Share IPD: No